CLINICAL TRIAL: NCT02709746
Title: Interventional, Randomised, Double-blind, Placebo-controlled, Active Reference (Fluoxetine), Fixed-dose Study of Vortioxetine in Paediatric Patients Aged 12 to 17 Years, With Major Depressive Disorder (MDD)
Brief Title: Active Reference (Fluoxetine) Fixed-dose Study of Vortioxetine in Paediatric Patients Aged 12 to 17 Years With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12710A; 2008-005354-20 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Depressive Disorder, Major
Keywords: paediatric patients
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vortioxetine 10 mg/day (Experimental)
  Interventions: Drug: Vortioxetine 10 mg/day
- Vortioxetine 20 mg/day (Experimental)
  Interventions: Drug: Vortioxetine 20 mg/day
- Fluoxetine 20 mg/day, (Active Comparator)
  Interventions: Drug: Fluoxetine 20 mg/day
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vortioxetine 10 mg/day — 10 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
  Other Names: Brintellix ®; Lu AA21004
  Arms: Vortioxetine 10 mg/day
Drug: Vortioxetine 20 mg/day — 20 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
  Other Names: Brintellix ®; Lu AA21004
  Arms: Vortioxetine 20 mg/day
Drug: Fluoxetine 20 mg/day — 20 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 10 mg/day. No dose increase will be allowed
  Arms: Fluoxetine 20 mg/day,
Other: Placebo — Encapsulated tablet
  Arms: Placebo

SUMMARY:
Evaluating the efficacy of vortioxetine 10 mg/day and 20 mg/day versus placebo on depressive symptoms in adolescents (age ≥12 and ≤17 years) with a DSM-5™ (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) diagnosis of Major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or female, aged ≥12 and ≤17 years at Screening (patients who turn 18 years during the study will be allowed to continue in the study).
* The patient has Major depressive disorder (MDD), diagnosed according to DSM-5™.
* The patient has a Children Depression Rating Scale - Revised (CDRS-R) total score ≥45 at the Screening Visit and at the Baseline.
* The patient has a Clinical Global Impression - Severity of Illness (CGI-S) score ≥4 at the Screening Visit and at the Baseline
* The patient has provided assent to participation and parent(s)/legal representative (s) signed the Informed Consent Form.

Exclusion Criteria:

* The patient has participated in a clinical study <30 days prior to the Screening Visit.

Other protocol defined inclusion and exclusion criteria may apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 784 (Actual)
Dates: Start 2016-05; Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (124):
- United States (42):
  - US1369, Dothan, Alabama
  - US1333, Tucson, Arizona
  - US1310, Little Rock, Arkansas
  - US1062, Costa Mesa, California
  - US1387, Downey, California
  - US1114, Escondido, California
  - US1118, Glendale, California
  - US1123, Imperial, California
  - US1160 Renew Behavioral Health, Inc., Long Beach, California
  - US1368, Orange, California
  - US1370, Panorama City, California
  - US1351, Wildomar, California
  - US1133, Washington D.C., District of Columbia
  - US1217, Gainesville, Florida
  - US1229, Orange City, Florida
  - US1009, Atlanta, Georgia
  - US1313, Marietta, Georgia
  - US1311, Naperville, Illinois
  - US1315, Naperville, Illinois
  - US1103, Oak Brook, Illinois
  - US1386, Wichita, Kansas
  - US1261, Lake Charles, Louisiana
  - US1015, Baltimore, Maryland
  - US1385 Ericksen Research And Development, Clinton, Mississippi
  - US1064, Creve Coeur, Missouri
  - US1314, O'Fallon, Missouri
  - US1266, Saint Charles, Missouri
  - US1312, Berlin, New Jersey
  - US1222, Princeton, New Jersey
  - US1317, New York, New York
  - US1171, Rochester, New York
  - US1190, Staten Island, New York
  - US1051, Cincinnati, Ohio
  - US1054, Cleveland, Ohio
  - US1334, Middleburg Heights, Ohio
  - US1323, Oklahoma City, Oklahoma
  - US1329, Oklahoma City, Oklahoma
  - US1328, Austin, Texas
  - US1320, Plano, Texas
  - US1162, San Antonio, Texas
  - US1308, Orem, Utah
  - US1309, Richmond, Virginia
- Bulgaria (2):
  - BG1023, Targovishte
  - BG1025, Varna
- Canada (2):
  - CA1036 University of Calgary, Calgary
  - CA1038, Toronto
- Colombia (4):
  - CO1003, Barranquilla
  - CO1001, Bello
  - CO1004, Bogotá
  - CO1002, Pereira
- Estonia (2):
  - EE1007, Tallinn
  - EE1015, Viljandi
- France (3):
  - FR1041, Douai
  - FR1017, Élancourt
  - FR1009, Nantes
- Germany (5):
  - DE1078, Freiburg im Breisgau
  - DE1034, Mainz
  - DE1077, Mannheim
  - DE1081, Maulbronn
  - DE1076, Tübingen
- Hungary (2):
  - HU1023, Budapest
  - HU1020, Gyula
- Italy (7):
  - IT1075, Cagliari
  - IT1073, Genova
  - IT1029, Messina
  - IT1068, Napoli
  - IT1074, Padua
  - IT1070, Pisa
  - IT1072 Osppedale Bambin gesu, Rome
- Latvia (4):
  - LV1002, Jelgava
  - LV1008, Liepāja
  - LV1009, Riga
  - LV1007, Sigulda
- Mexico (7):
  - MX1014, Culiacán
  - MX1011, Guadalajara
  - MX1013, Guadalajara
  - MX1022, Guadalajara
  - MX1023, Mazatlán
  - MX1003, Mexico City
  - MX1001, Nuevo León
- Poland (7):
  - PL1002, Bialystok
  - PL1050, Gdansk
  - PL1068, Kielce
  - PL1057, Lublin
  - PL1052, Poznan
  - PL1054, Wąbrzeźno
  - PL1051, Wroclaw
- Russia (14):
  - RU1009, Arkhangelsk
  - RU1059, Engel's
  - RU1046, Krasnodar
  - RU1011, Lipetsk
  - RU1004, Nizhny Novgorod
  - RU1010, Novosibirsk
  - RU1012, Rostov-on-Don
  - RU1044, Rostov-on-Don
  - RU1030, Saint Petersburg
  - RU1013, Saratov
  - RU1038, Saratov
  - RU1057, Tomsk
  - RU1048, Tonnel’nyy
  - RU1016, Yekaterinburg
- Serbia (5):
  - RS1006 Clinic of Neurology and Psychiatry for Children and Adolescents, Belgrade
  - RS1010, Belgrade
  - RS1011, Kragujevac
  - RS1003, Niš
  - RS1007, Novi Sad
- South Africa (3):
  - ZA1019, Cape Town
  - ZA1022, Randburg
  - ZA1023, Sandton
- South Korea (4):
  - KR1035, Cheonan
  - UA1037, Gyeongsang
  - KR1032, Seoul
  - KR1038, Seoul
- Spain (5):
  - ES1041, Alcorcón
  - ES1044, Madrid
  - ES1043, Pamplona
  - ES1018 Hospital de Sabadell, Sabadell
  - ES1040, Torremolinos
- Ukraine (4):
  - UA1002, Kyiv
  - UA1019, Odesa
  - UA1001, Poltava
  - UA1004, Ternopil
- United Kingdom (2):
  - GB1051, Glasgow
  - GB1047, Liverpool

REFERENCES:
- [Derived] Findling RL, DelBello MP, Zuddas A, Emslie GJ, Ettrup A, Petersen ML, Schmidt SN, Rosen M. Vortioxetine for Major Depressive Disorder in Adolescents: 12-Week Randomized, Placebo-Controlled, Fluoxetine-Referenced, Fixed-Dose Study. J Am Acad Child Adolesc Psychiatry. 2022 Sep;61(9):1106-1118.e2. doi: 10.1016/j.jaac.2022.01.004. Epub 2022 Jan 13. PMID 35033635

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who did not fulfil the randomization criteria for the Double-blind treatment (DBT) Period, were withdrawn from the study after the Single-blind treatment (SBT) period. Patients who fulfilled the randomization criteria for the DBT Period, continued into the DBT Period.
Groups:
- Single-blind Treatment, Placebo; DBT, Placebo: Placebo, encapsulated, orally
- DBT, Vortioxetine 10 mg: Vortioxetine 10 mg/day: 10 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
- DBT, Vortioxetine 20 mg: Vortioxetine 20 mg/day: 20 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
- DBT, Fluoxetine 20 mg: Fluoxetine 20 mg/day: 20 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 10 mg/day. No dose increase will be allowed
Period: Phase A (Single-blind Treatment Period)
Arm/Group | Single-blind Treatment, Placebo | DBT, Vortioxetine 10 mg | DBT, Vortioxetine 20 mg | DBT, Fluoxetine 20 mg | DBT, Placebo
Started | 784 | 0 | 0 | 0 | 0
Completed | 616 | 0 | 0 | 0 | 0
Not Completed | 168 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 0 | 0
Not completed — Not sepcified | 14 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 12 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0 | 0
Not completed — Enrolled not treated | 7 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0 | 0 | 0
Not completed — Do not fulfill rand criteria for DBT | 103 | 0 | 0 | 0 | 0
Period: Phase B (Double-blind Treatment Period)
Arm/Group | Single-blind Treatment, Placebo | DBT, Vortioxetine 10 mg | DBT, Vortioxetine 20 mg | DBT, Fluoxetine 20 mg | DBT, Placebo
Started | 0 | 147 | 162 | 153 | 154
Completed | 0 | 126 | 140 | 138 | 138
Not Completed | 0 | 21 | 22 | 15 | 16
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 2
Not completed — Other | 0 | 6 | 5 | 6 | 7
Not completed — Non-compliance with study drug | 0 | 1 | 4 | 1 | 0
Not completed — Lack of Efficacy | 0 | 3 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 4 | 8 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 2 | 1
Not completed — enrolled not treated | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Single-blind Treatment (SBT), Placebo: Single-blind treatment, Placebo (encapsulated, orally) and Brief Psychosocial Intervention (BPI) for 4 weeks
- DBT, Vortioxetine 10 mg: Eligible patients from SBT period (patients with incomplete improvement), will be randomly assigned (1:1:1:1) double-blind treatment in DBT Period, 8 weeks.
  Vortioxetine 10 mg/day, encapsulated tablets, orally.
- DBT, Vortioxetine 20 mg: Eligible patients from SBT period (patients with incomplete improvement), will be randomly assigned (1:1:1:1) double-blind treatment in DBT Period, 8 weeks.
  Vortioxetine 20 mg/day, encapsulated tablets, orally.
- DBT, Fluoxetine 20 mg: Eligible patients from SBT period (patients with incomplete improvement), will be randomly assigned (1:1:1:1) double-blind treatment in DBT Period, 8 weeks.
  Fluoxetine 20 mg/day, encapsulated tablets, orally.
- DBT, Placebo: Eligible patients from SBT period (patients with incomplete improvement), will be randomly assigned (1:1:1:1) double-blind treatment in DBT Period, 8 weeks.
  Placebo, encapsulated tablets, orally.
- Total: Total of all reporting groups
Arm/Group | Single-blind Treatment (SBT), Placebo | DBT, Vortioxetine 10 mg | DBT, Vortioxetine 20 mg | DBT, Fluoxetine 20 mg | DBT, Placebo | Total
Number analyzed (Participants) | 168 | 147 | 162 | 153 | 154 | 784
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.61) | 14.8 (1.66) | 14.5 (1.63) | 14.8 (1.60) | 14.6 (1.60) | 14.67 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 93 | 97 | 103 | 105 | 509
  Male | 57 | 54 | 65 | 50 | 49 | 275
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 4 | 2 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 37 | 19 | 19 | 20 | 22 | 117
  White | 108 | 108 | 110 | 112 | 106 | 544
  More than one race | 15 | 17 | 25 | 17 | 21 | 95
  Unknown or Not Reported | 4 | 3 | 4 | 2 | 1 | 14
CDRS-R total score at Enrolment [Least Squares Mean (Standard Deviation); unit: units on a scale] — The CDRS-R is a clinician-rated scale to measure the severity of depression of children and adolescents. The CDRS-R consists of 17 items: 14 items rate verbal observations, and three items rate nonverbal observations (tempo of language, hypoactivity, and nonverbal expression of depressed affect). Depression symptoms are rated on a 5-point scale from 1 to 5 for the verbal observations, and a 7-point scale from 1 to 7 for the nonverbal observations. The total score ranges from 17 (normal) to 113 (severe depression).
  units on a scale | 61.24 (10.00) | 64.82 (9.38) | 65.29 (9.73) | 64.06 (8.65) | 64.02 (8.96) | 63.85 (9.46)
CGI-S at Enrolment [Least Squares Mean (Standard Deviation); unit: units on a scale] — The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.82 (0.68) | 4.99 (0.77) | 5.00 (0.71) | 4.97 (0.68) | 4.92 (0.69) | 4.94 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Children Depression Rating Scale - Revised (CDRS-R) Total Score After Treatment
Description: The CDRS-R is a clinician-rated scale to measure the severity of depression of children and adolescents. The CDRS-R consists of 17 items: 14 items rate verbal observations, and three items rate nonverbal observations (tempo of language, hypoactivity, and nonverbal expression of depressed affect). Depression symptoms are rated on a 5-point scale from 1 to 5 for the verbal observations, and a 7-point scale from 1 to 7 for the nonverbal observations. The total score ranges from 17 (normal) to 113 (severe depression).
Time Frame: From Randomization to Week 8
Population: Double-blind treatment period
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Vortioxetine Average (Avg. VOR): patients are randomized to one of four treatments.
  Avg.- VOR is a calculation based on the treatment estimates from VOR 10 mg and VOR 20 mg.
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo | Vortioxetine Average (Avg. VOR)
Number analyzed (Participants) | 126 | 139 | 137 | 137 | 265
units on a scale | -17.09 (1.27) | -18.94 (1.22) | -21.95 (1.23) | -18.22 (1.22) | -18.01 (0.98)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg/Day vs Placebo; Test type: Superiority; p = 0.4702, Mixed Model Repeated Analysis; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-1.94 to 4.2]
Statistical Analysis 2: Comparison: Vortioxetine 20 mg/Day vs Placebo; Test type: Superiority; p = 0.6373, Mixed Model Repeated Analysis; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-3.71 to 2.27]
Statistical Analysis 3: Comparison: Fluoxetine 20 mg/Day, vs Placebo; Test type: Superiority; p = 0.0152, Mixed Model Repeated Analysis; Mean Difference (Final Values) = -3.73, 95% CI 2-sided [-6.74 to -0.72]
Statistical Analysis 4: Comparison: Placebo vs Vortioxetine Average (Avg. VOR); Test type: Superiority; p = 0.8778, Mixed Model Repeated Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-2.41 to 2.82]

2. Secondary Outcome: Change in CDRS-R Total Score During Treatment (at Week 2)
Description: The CDRS-R is a clinician-rated scale to measure the severity of depression of children and adolescents. The CDRS-R consists of 17 items: 14 items rate verbal observations, and three items rate nonverbal observations (tempo of language, hypoactivity, and nonverbal expression of depressed affect). Depression symptoms are rated on a 5-point scale from 1 to 5 for the verbal observations, and a 7-point scale from 1 to 7 for the nonverbal observations. The total score ranges from 17 (normal) to 113 (severe depression).Children and parents answer separately. Rater judges and selects 'Best'.
Time Frame: At week 2
Population: Double-blind treatment period. There where overall numbers of participants analyzed are not consistent with numbers provided in the participant flow can be due to particpant flow module total number of patients also includes patients that were enrolled but not treated and other reasons of discontinuation from the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 145 | 158 | 150 | 153
units on a scale | -9.58 (1.02) | -10.15 (0.99) | -10.34 (1.00) | -8.83 (0.98)

3. Secondary Outcome: Change in CDRS-R Total Score During Treatment (at Week 4)
Description: as for outcome 1
Time Frame: At week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 137 | 153 | 145 | 149
units on a scale | -14.32 (1.14) | -15.03 (1.10) | -16.25 (1.11) | -13.71 (1.09)

4. Secondary Outcome: Change in CDRS-R Total Score During Treatment (at Week 6)
Description: as for outcome 1
Time Frame: At week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 127 | 145 | 143 | 142
units on a scale | -15.43 (1.24) | -17.78 (1.19) | -19.20 (1.2) | -16.71 (1.19)

5. Secondary Outcome: Change in CDRS-R Mood Score
Description: Change in Children Depression Rating Scale - Revised (CDRS-R) Mood. The CDRS-R has been widely used for the evaluation of children and adolescents with major depressive disorder (MDD). The CDRS-R total score is the sum of the responses to 17 items. Each item is graded on a 5- or 7-point scale. Mood is one of four subscores defined in the CDRS-R: sum of items 8, 11, 14, 15; score range 4 to 28. The highest possible score indicates the most severe measure of depression.
Time Frame: From randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -5.05 (0.40) | -5.47 (0.38) | -6.53 (0.38) | -5.32 (0.38)

6. Secondary Outcome: Change in CDRS-R Somatic Score
Description: Change in Children Depression Rating Scale - Revised (CDRS-R): Somatic. The CDRS-R has been widely used for the evaluation of children and adolescents with major depressive disorder (MDD). The CDRS-R total score is the sum of the responses to 17 items. Each item is graded on a 5- or 7-point scale. Somatic is one of four subscores defined in the CDRS-R: sum of items 4, 5, 6, 7, 16, 17; score ranges from 6 to 36. The highest possible score indicates the most severe measure of depression.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -5.63 (0.46) | -6.03 (0.44) | -6.79 (0.45) | -5.78 (0.44)

7. Secondary Outcome: Change in CDRS-R Subjective Score
Description: Change in Children Depression Rating Scale - Revised (CDRS-R): Subjective. The CDRS-R has been widely used for the evaluation of children and adolescents with major depressive disorder (MDD). The CDRS-R total score is the sum of the responses to 17 items. Each item is graded on a 5- or 7-point scale. Subjective is one of four subscores defined in the CDRS-R: sum of items 9, 10, 12, 13; score ranges from 4 to 28. The highest possible score indicates the most severe measure of depression.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -2.41 (0.22) | -2.63 (0.21) | -3.23 (0.21) | -2.66 (0.21)

8. Secondary Outcome: Change in CDRS-R Behaviour Score
Description: Change in Children Depression Rating Scale - Revised (CDRS-R): Behaviour. The CDRS-R has been widely used for the evaluation of children and adolescents with major depressive disorder (MDD). The CDRS-R total score is the sum of the responses to 17 items. Each item is graded on a 5- or 7-point scale. behaviour is one of four subscores defined in the CDRS-R:sum of items 1, 2, 3; score ranges from 3 to 21. The highest possible score indicates the most severe measure of depression.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -4.32 (0.38) | -4.90 (0.36) | -5.52 (0.37) | -4.73 (0.36)

9. Secondary Outcome: CDRS-R Response
Description: Children Depression Rating Scale - Response: defined as a >= 50% decrease in CDRS-R total score, calculated as (change from baseline [Randomization])/(baseline value - 17).
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
Participants | 53 | 60 | 68 | 49

10. Secondary Outcome: CDRS-R Remission
Description: Remission is defined as a CDRS-R total score <= 28.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
Participants | 21 | 24 | 32 | 20

11. Secondary Outcome: Change in General Behaviour Inventory (GBI) Depression Sub Scale Score Assessed by the Parents
Description: Using the 10-item depression subscale, assessed by parent (PGBI-10D). Change from randomization to Week 8 in GBI Total Parent/Guardian Version Depression score. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale completed by parent/guardian. Symptoms rated on 4-point Likert scale from 0 (never/hardly ever) to 3 (often/almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: From randomization to week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -6.23 (0.56) | -6.48 (0.54) | -8.00 (0.54) | -6.62 (0.53)

12. Secondary Outcome: Change General Behaviour Inventory (GBI) Depression Subscale Score Assessed by the Child
Description: The GBI 10-item mania scale is a parent- and subject-rated scale designed to screen for manic symptoms in children and adolescents. The 10 items are rated on a scale from 0 (never or hardly ever) to 3 (very often or almost constantly). The total score ranges from 0 to 30 points, with high scores indicating greater pathology.
Time Frame: From randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -5.48 (0.61) | -5.55 (0.59) | -6.30 (0.59) | -6.03 (0.58)

13. Secondary Outcome: Parent Global Assessment-Global Improvement (PGA) Score
Description: The PGA is a parent-rated variation of the CGI-I to evaluate the severity of the child's symptoms. The PGA reflects assessments of change from Baseline symptoms using a 7 point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 125 | 139 | 137 | 137
units on a scale | 2.80 (0.10) | 2.74 (0.09) | 2.49 (0.09) | 2.72 (0.09)

14. Secondary Outcome: Change in Symbol Digit Modalities Test (SDMT)
Description: The Symbol Digit Modalities Test (SDMT) is a cognitive test designed to assess speed of performance requiring visual perception, spatial decision-making and psychomotor skills. The SDMT consists of 110 geometric symbols that the patient has to substitute with a corresponding digit in a 90-second period. Each correct digit is counted, and the total score ranges from 0 (less than normal functioning) to 110 (greater than normal functioning).
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 125 | 140 | 138 | 137
units on a scale | 3.75 (1.02) | 2.64 (0.98) | 2.69 (0.98) | 2.41 (0.97)

15. Secondary Outcome: Change in Clinical Global Impression Severity of Illness (CGI-S) Score
Description: The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
units on a scale | -1.23 (0.10) | -1.38 (0.10) | -1.59 (0.10) | -1.21 (0.10)

16. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score
Description: The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 125 | 139 | 137 | 137
units on a scale | 2.81 (0.10) | 2.69 (0.09) | 2.50 (0.09) | 2.73 (0.09)

17. Secondary Outcome: CGI-S Remission
Description: Remission defined as CGI-S score of 1 or 2.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 139 | 137 | 137
Participants | 26 | 33 | 36 | 24

18. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS) Score
Description: The Children's Global Assessment Score (CGAS) is a rating scale which measures psychological, social and school functioning for children. The CGAS is a clinician-rated global scale to measure the lowest level of functioning for a child (4 to 16 years) during a specified time period. The CGAS contains behaviourally oriented descriptors at each anchor point that depict behaviours and life situations applicable to a child. The items range in value from 1 (most functionally impaired child) to 100 (the healthiest). A total score above 70 indicates normal function.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 126 | 140 | 138 | 137
units on a scale | 12.24 (1.25) | 13.89 (1.20) | 16.43 (1.20) | 14.52 (1.19)

19. Secondary Outcome: Change in Pediatric Quality of Life Inventory (PedsQL) Visual Analogue Scales (VAS): Afraid or Scared (Anxiety) Score
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue and pain using visual analogue scales. The functionality for each domain is measured on a 10 cm line with a happy face at one end and a sad face at the other (0-10 points). The patients are asked to mark on the line how they feel. A lower value represents a better outcome.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -0.47 (0.19) | -0.76 (0.18) | -0.78 (0.18) | -0.71 (0.18)

20. Secondary Outcome: Change in PedsQL VAS: Sad or Blue (Sadness) Score
Description: as for outcome 19
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -1.90 (0.26) | -1.71 (0.25) | -2.45 (0.25) | -2.12 (0.24)

21. Secondary Outcome: Change in PedsQL VAS: Angry Score
Description: as for outcome 19
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -0.51 (0.23) | -0.70 (0.23) | -1.01 (0.23) | -0.59 (0.23)

22. Secondary Outcome: Change in PedsQL VAS: Worry Score
Description: as for outcome 19
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -0.96 (0.25) | -1.17 (0.24) | -0.91 (0.24) | -1.33 (0.24)

23. Secondary Outcome: Change in PedsQL VAS: Tired (Fatigue) Score
Description: as for outcome 19
Time Frame: From Randomization to week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -1.18 (0.29) | -1.40 (0.28) | -1.55 (0.28) | -1.27 (0.28)

24. Secondary Outcome: Change in PedsQL VAS: Pain or Hurt Score
Description: as for outcome 19
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -1.12 (0.22) | -0.97 (0.21) | -0.83 (0.21) | -0.76 (0.21)

25. Secondary Outcome: Change in PedsQL VAS Total Average Score
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL™ VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue, and pain using visual analogue scales. The functionality for each domain is measured on a 10cm line with a happy face at one end and a sad face at the other (0-10 points). The patients are asked to mark on the line how they feel. The total score is the average of all 6 items. A lower value represents a better outcome.
Time Frame: From Randomization to week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -1.00 (0.17) | -1.13 (0.16) | -1.33 (0.16) | -1.14 (0.16)

26. Secondary Outcome: Change in PedsQL Emotional Distress Summary Average Score
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue and pain using visual analogue scales. The functionality for each domain is measured on a 10 cm line with a happy face at one end and a sad face at the other (0-10 points). The patients are asked to mark on the line how they feel. The average emotional distress summary score is the mean of the anxiety, sadness, anger, and worry items. A lower value represents a better outcome.
Time Frame: From Randomization to week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 124 | 140 | 138 | 137
units on a scale | -0.93 (0.18) | -1.09 (0.17) | -1.33 (0.17) | -1.18 (0.17)

27. Secondary Outcome: Change in Paediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Total Scores
Description: PQ-LES-Q total score (items 1 to 14). The PQ-LES-Q is a patient-rated scale designed to assess satisfaction with life. It is an adaptation of the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), which is used to measure quality of life in adults. The PQ LES Q consist of 15 items, item 1-14 assess the degree of satisfaction experienced by subjects in various areas of daily functioning (and item 15 allows subjects to summarize their experience in a global rating). Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good). The total score range of item 1-14 (this outcome measurement) is 14 to 70, with higher scores indicating greater satisfaction.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 125 | 140 | 137 | 137
units on a scale | 7.62 (0.97) | 7.56 (0.93) | 9.26 (0.94) | 7.06 (0.92)

28. Secondary Outcome: Change in PQ-LES-Q Overall Score
Description: PQ-LES-Q overall evaluation score (item 15). The PQ-LES-Q is a patient-rated scale designed to assess satisfaction with life. It is an adaptation of the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), which is used to measure quality of life in adults. The PQ-LES-Q consist of 15 items, item 1-14 assess the degree of satisfaction experienced by subjects in various areas of daily functioning and item 15 allows subjects to summarize their experience in a global rating (this outcome measurement). Item 15 is rated on a 5-point scale from 1 (very poor) to 5 (very good).
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg/Day | Vortioxetine 20 mg/Day | Fluoxetine 20 mg/Day, | Placebo
Number analyzed (Participants) | 125 | 140 | 137 | 137
units on a scale | 0.54 (0.08) | 0.43 (0.08) | 0.67 (0.08) | 0.51 (0.08)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: There where the total numbers of participants at risk are not onsistent with numbers provided in the particpant flow module is due that patients that were enrolled but not treated are included in the total number in the participant flow module.
Groups:
- SBT, Placebo: Patients not randomized to DBT period
- DBT, Fluoxetine 20 mg: Vortioxetine 20 mg/day: 10 mg/day, encapsulated tablet (with addition of lower initial dose levels). Based on tolerability the dose may be reduced by 10 mg/day. No dose increase will be allowed
- DBT, Placebo: Placebo, encapsulated tablet, orally
Arm/Group | SBT, Placebo | DBT, Vortioxetine 10 mg | DBT, Vortioxetine 20 mg | DBT, Fluoxetine 20 mg | DBT, Placebo
All-Cause Mortality (participants affected / at risk) | 0/777 | 0/147 | 0/161 | 0/153 | 0/154
Serious Adverse Events (participants affected / at risk) | 13/777 | 4/147 | 7/161 | 3/153 | 1/154
Other Adverse Events (participants affected / at risk) | 128/777 | 47/147 | 57/161 | 40/153 | 30/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBT, Placebo (N=777) | DBT, Vortioxetine 10 mg (N=147) | DBT, Vortioxetine 20 mg (N=161) | DBT, Fluoxetine 20 mg (N=153) | DBT, Placebo (N=154)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 6 (6) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBT, Placebo (N=777) | DBT, Vortioxetine 10 mg (N=147) | DBT, Vortioxetine 20 mg (N=161) | DBT, Fluoxetine 20 mg (N=153) | DBT, Placebo (N=154)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 5 (5) | 9 (10) | 7 (11) | 5 (5)
Nausea (Gastrointestinal disorders) | 28 (31) | 21 (23) | 31 (48) | 10 (16) | 7 (9)
Vomiting (Gastrointestinal disorders) | 13 (13) | 7 (7) | 15 (20) | 8 (10) | 1 (1)
Nasopharyngitis (Infections and infestations) | 26 (28) | 6 (7) | 10 (11) | 10 (12) | 5 (7)
Dizziness (Nervous system disorders) | 21 (23) | 11 (14) | 7 (7) | 6 (8) | 5 (6)
Headache (Nervous system disorders) | 65 (85) | 23 (37) | 20 (46) | 10 (16) | 12 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT02709746/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02709746/SAP_001.pdf